CLINICAL TRIAL: NCT04503382
Title: An Exploratory Study of the Impact of Kindness Videos in Health Care Settings
Brief Title: Impact of Kindness Videos in Health Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Envision Kindness Inc (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK-002
Record Dates: First submitted 2020-07-28; First posted 2020-08-07 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Altruism; Behavior; Emotions
Keywords: kindness; behavior; altruism; emotions; generosity
MeSH Terms: conditions — Altruism; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kindness media (Experimental): Short videos of kindness media. As part of a program entitled EnSpire®, this media consists of short videos that display acts of kindness and compassion that are edited together into a single reel.
  Interventions: Other: Kindness Media
- Standard television (Active Comparator): Children's commercial programming--as the control condition, participants watched commercial children's programming such as Disney, Nickelodeon, etc.
  Interventions: Other: Kindness Media

INTERVENTIONS:
Other: Kindness Media — As described above, the intervention is a series of short videos that display acts of kindness or ideas about kindness. These videos are edited together into one reel that was 8 minutes long.
  Other Names: EnSpire®

SUMMARY:
This study builds on earlier work assessing the impact of kindness media on viewers' emotional responses. Using images of kindness and connection, as well as other content, we will test its impact on emotions and behavior in the field. The setting is in healthcare, specifically a pediatric dental clinic. Using simple scales, participants anonymously rate themselves on a variety of emotions, watch a television for 8 minutes, and then complete the self-assessment. An honorarium is provided for participation.

DETAILED DESCRIPTION:
The present study builds on the earlier work with a focused application of inspiring content in health care settings. It is well described that health care providers, including doctors, nurses, and other staff members) have high rates of burnout, depression, and suicide-approximately twice that of the general population. In addition to the lower quality of life for the individual health care provider, this burnout problem has consequences for the patient, including heightened number of medical errors.

Patients, of course, also have significant stressors in their lives. Perhaps, those center on health-related issues, or are more general in nature. In the general population, it is known that anxiety, perceived stress, opiate abuse, and suicide are all rising.

From the patients' perspective, it is important to encourage them to adapt behaviors and attitudes that will benefit themselves as well as others. It has been shown that being kind and compassionate can yield positive impacts on health: people who volunteer regularly, for example, have death rates 20-40% lower than those who do not. Another facet of inducing kindness and compassion is kindness towards oneself. In health care settings, behavioral modification is very challenging. One way to rethink that approach is teaching and illustrating to patients how kindness to oneself is a necessity. Kindness to oneself encompasses following physician instructions as well as general health practice. By providing inspiring visual content to both patients and providers, it is believed that at least additive if not synergistic interaction will occur with simultaneous promotion of kindness, compassion, joy and love for both groups.

To date, multiple publications have pointed to the observation that various types of media can inspire viewers such that they are "moved" or "touched" or "elevated." Most of these studies have focused on the use of single films from several minutes long to full length feature films.

Much of the above cited research has been done in a laboratory or structured research setting. While very valuable, this research plan focuses on a "real world" setting, i.e., with patients and practitioners at the source in their work environments. The first step is to measure responses from both providers and patients.

C. Objectives

1. Quantify the response to videos depicting kindness, compassion, connection, joy, and love for both patients (or caregivers) and for health care staff.
2. Compare these responses to the standard content that the site uses.
3. Determine the impact of these videos on a measure of generosity.
4. Obtain qualitative feedback on the content in the effort to improve the content.

D. Hypothesis

1. Kindness media both moves and provides a significant lift in emotional state for both sets of viewers (providers and patients).
2. Compared to what is usually shown, kindness media has significant impact on emotional state.
3. Viewers will prefer to see more kindness media upon future visits.

Design:

Open, randomized, comparator-controlled study of kindness media versus commercial media on emotions and behavior. Parents and staff of the clinic are recruited as participants. Surveys with self-ratings are completed before and then after watching either kindness media or commercial (standard) children's media for 8 minutes.

ELIGIBILITY:
Inclusion Criteria:

- Ability to give consent and complete forms

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Emotional responses | immediately after intervention
  Set of questions regarding self-assessed emotional states including happiness, feeling calm, grateful, compassionate, optimistic, sad, irritated, or anxious. Scored 1-5 with "1" = not at all and "5"= a lot.

SECONDARY OUTCOMES:
Number of participants who donated | Immediately after intervention
  Measurement of donation--participants are asked whether or not they would be willing to donate to a family in need. The number of donations in each intervention group is counted.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Dental Associates of New London County, New London, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No